CLINICAL TRIAL: NCT05049200
Title: Epidemiology of Weaning From Invasive Mechanical Ventilation in COVID-19. Observational and Multicenter Study.
Brief Title: Characteristics of Weaning From Mechanical Ventilation in COVID-19
Acronym: CovWean
Status: Completed | Type: Observational
Sponsor: Sanatorio Anchorena San Martin (Other)
Responsible Party: Principal Investigator, Matias Accoce, HEAD OF RESPIRATORY THERAPY, Sanatorio Anchorena San Martin
Other Study IDs: 15/16
Record Dates: First submitted 2021-09-16; First posted 2021-09-20 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Respiration, Artificial; COVID-19
Keywords: Respiration, Artificial; Ventilator Weaning; Airway Extubation; COVID-19
MeSH Terms: conditions — Respiratory Aspiration; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This report is a multicenter, observational, analytical and prospective study. The objective was to describe the weaning of mechanical ventilation in patients with SARS-CoV-2 and the clinical results according to the different types of weaning.

DETAILED DESCRIPTION:
This report is a multicenter, observational, analytical and prospective study.

Patients older than 18 years with a diagnosis of COVID-19 by PCR + and who required invasive VM for more than 12 hours from April 1 to August 30, 2020 were included. Subjects admitted to pediatric ICUs and in the recovery room were excluded. Patients who were readmitted and required a new cycle of MV after having been successfully weaned and released from the hospital were also excluded. All patients with data loss greater than 10% in variables considered clinically relevant were eliminated.

The weaning process from mechanical ventilation in each patient was classified by two strategies:

Definition of critical care medicine consensus conference published (2007) in:

Simple weaning: Patients successfully extubated after the first weaning attempt.

Difficult weaning: Patients who fail the first weaning attempt and require up to three spontaneous breathing trials or up to 7 days from the first spontaneous breathing trial to achieve a successful weaning.

Prolonged weaning: Patients who fail at least three weaning attempts or require more than 7 days after the first spontaneous breathing trial.

Definition of WIND study:

Group 0 ("no weaning"), made up of patients who never experienced any attempt to wean.

Group 1 (short weaning): the first attempt resulted in the completion of the weaning process in 1 day (successful weaning or early death).

Group 2 (difficult weaning): weaning was completed after more than 1 day but less than 1 week after the first attempt (successful weaning or death).

Group 3 (prolonged weaning): weaning is not yet completed 7 days after the first attempt (due to successful weaning or death).

The first attempt at weaning in intubated patients was considered as the performance of a spontaneous breathing trial with or without extubation, or extubation with or without SBT. In tracheostomized patients, the first period of spontaneous breathing (without ventilatory support) of at least 24 hours duration was considered as the first weaning attempt.

Weaning success was considered when death or re-intubation did not occur after extubation within 7 days or until discharge from the ICU (whichever occurs first), whether or not non-invasive ventilatory support was used. In tracheostomized patients, weaning was considered successful upon reaching seven consecutive days of spontaneous ventilation without ventilatory support or discharge from the ICU, whichever occurs first. [24]

The data were collected by the principal investigator of each center, or by one of the members of the work team designated for the study, preferably between 8:00 am and 11:00 am, recorded on paper sheets and dumped into a database " online "designed in REDCap (Research Electronic Data Capture) with software installed in the Centro del Parque clinic, Buenos Aires, Argentina, guaranteeing the protection and confidentiality of the data in accordance with the Declaration of Helsinki. Data were acquired from the moment of admission to the ICU (once the inclusion criteria and the absence of exclusion criteria had been met) and during the entire follow-up period. All members of the research group provided advice and support through direct telephone contact / e-mail specifically originated for the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COVID-19 by PCR +
* Invasive mechanical ventilation for more than 12 hours

Exclusion Criteria:

* Subjects admitted to pediatric ICUs and surgery recovery room.
* Patients who were readmitted and required a new cycle of invasive mechanical ventilation after having been successfully weaned and released from the hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of COVID-19 by PCR + and who required invasive mechanical ventilation for more than 12 hours were included.
Sampling Method: Non-Probability Sample
Enrollment: 326 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
weaning rate | on day 28
  percentage of successfully weaned patients
weaning classification | on day 28
  number of spontaneous breathing tests and days from first spontaneous breathing test to success or death

SECONDARY OUTCOMES:
mechanical ventilation days | on day 28
  duration of invasive mechanical ventilation
length of ICU stay | on day 28
  days of hospitalization in ICU

CONTACTS AND LOCATIONS:
Locations (2):
- Argentina (2):
  - Matias Accoce, Pereyra, Buenos Aires
  - Sanatorio Anchorena de San Martin, San Martín, Buenos Aires

REFERENCES:
- [Result] Ranzani OT, Bastos LSL, Gelli JGM, Marchesi JF, Baiao F, Hamacher S, Bozza FA. Characterisation of the first 250,000 hospital admissions for COVID-19 in Brazil: a retrospective analysis of nationwide data. Lancet Respir Med. 2021 Apr;9(4):407-418. doi: 10.1016/S2213-2600(20)30560-9. Epub 2021 Jan 15. PMID 33460571
- [Result] Estenssoro E, Loudet CI, Rios FG, Kanoore Edul VS, Plotnikow G, Andrian M, Romero I, Piezny D, Bezzi M, Mandich V, Groer C, Torres S, Orlandi C, Rubatto Birri PN, Valenti MF, Cunto E, Saenz MG, Tiribelli N, Aphalo V, Reina R, Dubin A; SATI-COVID-19 Study Group. Clinical characteristics and outcomes of invasively ventilated patients with COVID-19 in Argentina (SATICOVID): a prospective, multicentre cohort study. Lancet Respir Med. 2021 Sep;9(9):989-998. doi: 10.1016/S2213-2600(21)00229-0. Epub 2021 Jul 2. PMID 34224674
- [Result] Grasselli G, Zangrillo A, Zanella A, Antonelli M, Cabrini L, Castelli A, Cereda D, Coluccello A, Foti G, Fumagalli R, Iotti G, Latronico N, Lorini L, Merler S, Natalini G, Piatti A, Ranieri MV, Scandroglio AM, Storti E, Cecconi M, Pesenti A; COVID-19 Lombardy ICU Network. Baseline Characteristics and Outcomes of 1591 Patients Infected With SARS-CoV-2 Admitted to ICUs of the Lombardy Region, Italy. JAMA. 2020 Apr 28;323(16):1574-1581. doi: 10.1001/jama.2020.5394. PMID 32250385
- [Result] Karagiannidis C, Mostert C, Hentschker C, Voshaar T, Malzahn J, Schillinger G, Klauber J, Janssens U, Marx G, Weber-Carstens S, Kluge S, Pfeifer M, Grabenhenrich L, Welte T, Busse R. Case characteristics, resource use, and outcomes of 10 021 patients with COVID-19 admitted to 920 German hospitals: an observational study. Lancet Respir Med. 2020 Sep;8(9):853-862. doi: 10.1016/S2213-2600(20)30316-7. Epub 2020 Jul 28. PMID 32735842
- [Result] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337
- [Result] Esteban A, Frutos-Vivar F, Muriel A, Ferguson ND, Penuelas O, Abraira V, Raymondos K, Rios F, Nin N, Apezteguia C, Violi DA, Thille AW, Brochard L, Gonzalez M, Villagomez AJ, Hurtado J, Davies AR, Du B, Maggiore SM, Pelosi P, Soto L, Tomicic V, D'Empaire G, Matamis D, Abroug F, Moreno RP, Soares MA, Arabi Y, Sandi F, Jibaja M, Amin P, Koh Y, Kuiper MA, Bulow HH, Zeggwagh AA, Anzueto A. Evolution of mortality over time in patients receiving mechanical ventilation. Am J Respir Crit Care Med. 2013 Jul 15;188(2):220-30. doi: 10.1164/rccm.201212-2169OC. PMID 23631814
- [Result] Kress JP, Pohlman AS, O'Connor MF, Hall JB. Daily interruption of sedative infusions in critically ill patients undergoing mechanical ventilation. N Engl J Med. 2000 May 18;342(20):1471-7. doi: 10.1056/NEJM200005183422002. PMID 10816184
- [Result] Girard TD, Kress JP, Fuchs BD, Thomason JW, Schweickert WD, Pun BT, Taichman DB, Dunn JG, Pohlman AS, Kinniry PA, Jackson JC, Canonico AE, Light RW, Shintani AK, Thompson JL, Gordon SM, Hall JB, Dittus RS, Bernard GR, Ely EW. Efficacy and safety of a paired sedation and ventilator weaning protocol for mechanically ventilated patients in intensive care (Awakening and Breathing Controlled trial): a randomised controlled trial. Lancet. 2008 Jan 12;371(9607):126-34. doi: 10.1016/S0140-6736(08)60105-1. PMID 18191684
- [Result] Morandi A, Brummel NE, Ely EW. Sedation, delirium and mechanical ventilation: the 'ABCDE' approach. Curr Opin Crit Care. 2011 Feb;17(1):43-9. doi: 10.1097/MCC.0b013e3283427243. PMID 21169829
- [Result] Vincent JL, Shehabi Y, Walsh TS, Pandharipande PP, Ball JA, Spronk P, Longrois D, Strom T, Conti G, Funk GC, Badenes R, Mantz J, Spies C, Takala J. Comfort and patient-centred care without excessive sedation: the eCASH concept. Intensive Care Med. 2016 Jun;42(6):962-71. doi: 10.1007/s00134-016-4297-4. Epub 2016 Apr 13. PMID 27075762
- [Result] Balas MC, Vasilevskis EE, Olsen KM, Schmid KK, Shostrom V, Cohen MZ, Peitz G, Gannon DE, Sisson J, Sullivan J, Stothert JC, Lazure J, Nuss SL, Jawa RS, Freihaut F, Ely EW, Burke WJ. Effectiveness and safety of the awakening and breathing coordination, delirium monitoring/management, and early exercise/mobility bundle. Crit Care Med. 2014 May;42(5):1024-36. doi: 10.1097/CCM.0000000000000129. PMID 24394627
- [Result] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Result] Liu K, Nakamura K, Katsukawa H, Elhadi M, Nydahl P, Ely EW, Kudchadkar SR, Takahashi K, Inoue S, Lefor AK, Kesecioglu J, Nishida O. ABCDEF Bundle and Supportive ICU Practices for Patients With Coronavirus Disease 2019 Infection: An International Point Prevalence Study. Crit Care Explor. 2021 Mar 12;3(3):e0353. doi: 10.1097/CCE.0000000000000353. eCollection 2021 Mar. PMID 33786432
- [Result] Ackermann M, Verleden SE, Kuehnel M, Haverich A, Welte T, Laenger F, Vanstapel A, Werlein C, Stark H, Tzankov A, Li WW, Li VW, Mentzer SJ, Jonigk D. Pulmonary Vascular Endothelialitis, Thrombosis, and Angiogenesis in Covid-19. N Engl J Med. 2020 Jul 9;383(2):120-128. doi: 10.1056/NEJMoa2015432. Epub 2020 May 21. PMID 32437596
- [Result] Marini JJ, Gattinoni L. Management of COVID-19 Respiratory Distress. JAMA. 2020 Jun 9;323(22):2329-2330. doi: 10.1001/jama.2020.6825. No abstract available. PMID 32329799
- [Result] Robba C, Battaglini D, Ball L, Patroniti N, Loconte M, Brunetti I, Vena A, Giacobbe DR, Bassetti M, Rocco PRM, Pelosi P. Distinct phenotypes require distinct respiratory management strategies in severe COVID-19. Respir Physiol Neurobiol. 2020 Aug;279:103455. doi: 10.1016/j.resp.2020.103455. Epub 2020 May 11. PMID 32437877
- [Result] Grasselli G, Tonetti T, Protti A, Langer T, Girardis M, Bellani G, Laffey J, Carrafiello G, Carsana L, Rizzuto C, Zanella A, Scaravilli V, Pizzilli G, Grieco DL, Di Meglio L, de Pascale G, Lanza E, Monteduro F, Zompatori M, Filippini C, Locatelli F, Cecconi M, Fumagalli R, Nava S, Vincent JL, Antonelli M, Slutsky AS, Pesenti A, Ranieri VM; collaborators. Pathophysiology of COVID-19-associated acute respiratory distress syndrome: a multicentre prospective observational study. Lancet Respir Med. 2020 Dec;8(12):1201-1208. doi: 10.1016/S2213-2600(20)30370-2. Epub 2020 Aug 27. PMID 32861276
- [Result] Gupta A, Madhavan MV, Sehgal K, Nair N, Mahajan S, Sehrawat TS, Bikdeli B, Ahluwalia N, Ausiello JC, Wan EY, Freedberg DE, Kirtane AJ, Parikh SA, Maurer MS, Nordvig AS, Accili D, Bathon JM, Mohan S, Bauer KA, Leon MB, Krumholz HM, Uriel N, Mehra MR, Elkind MSV, Stone GW, Schwartz A, Ho DD, Bilezikian JP, Landry DW. Extrapulmonary manifestations of COVID-19. Nat Med. 2020 Jul;26(7):1017-1032. doi: 10.1038/s41591-020-0968-3. Epub 2020 Jul 10. PMID 32651579
- [Result] Ionescu F, Zimmer MS, Petrescu I, Castillo E, Bozyk P, Abbas A, Abplanalp L, Dogra S, Nair GB. Extubation Failure in Critically Ill COVID-19 Patients: Risk Factors and Impact on In-Hospital Mortality. J Intensive Care Med. 2021 Sep;36(9):1018-1024. doi: 10.1177/08850666211020281. Epub 2021 Jun 2. PMID 34074160
- [Result] Cuschieri S. The STROBE guidelines. Saudi J Anaesth. 2019 Apr;13(Suppl 1):S31-S34. doi: 10.4103/sja.SJA_543_18. PMID 30930717
- [Result] Boles JM, Bion J, Connors A, Herridge M, Marsh B, Melot C, Pearl R, Silverman H, Stanchina M, Vieillard-Baron A, Welte T. Weaning from mechanical ventilation. Eur Respir J. 2007 May;29(5):1033-56. doi: 10.1183/09031936.00010206. PMID 17470624
- [Result] Beduneau G, Pham T, Schortgen F, Piquilloud L, Zogheib E, Jonas M, Grelon F, Runge I, Nicolas Terzi, Grange S, Barberet G, Guitard PG, Frat JP, Constan A, Chretien JM, Mancebo J, Mercat A, Richard JM, Brochard L; WIND (Weaning according to a New Definition) Study Group and the REVA (Reseau Europeen de Recherche en Ventilation Artificielle) Network double dagger. Epidemiology of Weaning Outcome according to a New Definition. The WIND Study. Am J Respir Crit Care Med. 2017 Mar 15;195(6):772-783. doi: 10.1164/rccm.201602-0320OC. PMID 27626706
- [Result] Righetti RF, Onoue MA, Politi FVA, Teixeira DT, Souza PN, Kondo CS, Moderno EV, Moraes IG, Maida ALV, Pastore Junior L, Silva FD, Brito CMM, Baia WRM, Yamaguti WP. Physiotherapy Care of Patients with Coronavirus Disease 2019 (COVID-19) - A Brazilian Experience. Clinics (Sao Paulo). 2020 Jun 22;75:e2017. doi: 10.6061/clinics/2020/e2017. eCollection 2020. PMID 32578825
- [Result] Kangas-Dick AW, Swearingen B, Wan E, Chawla K, Wiesel O. Safe extubation during the COVID-19 pandemic. Respir Med. 2020 Aug-Sep;170:106038. doi: 10.1016/j.rmed.2020.106038. Epub 2020 May 23. PMID 32469731
- [Result] Ouellette DR, Patel S, Girard TD, Morris PE, Schmidt GA, Truwit JD, Alhazzani W, Burns SM, Epstein SK, Esteban A, Fan E, Ferrer M, Fraser GL, Gong MN, Hough CL, Mehta S, Nanchal R, Pawlik AJ, Schweickert WD, Sessler CN, Strom T, Kress JP. Liberation From Mechanical Ventilation in Critically Ill Adults: An Official American College of Chest Physicians/American Thoracic Society Clinical Practice Guideline: Inspiratory Pressure Augmentation During Spontaneous Breathing Trials, Protocols Minimizing Sedation, and Noninvasive Ventilation Immediately After Extubation. Chest. 2017 Jan;151(1):166-180. doi: 10.1016/j.chest.2016.10.036. Epub 2016 Nov 3. PMID 27818331
- [Result] Cabello B, Thille AW, Roche-Campo F, Brochard L, Gomez FJ, Mancebo J. Physiological comparison of three spontaneous breathing trials in difficult-to-wean patients. Intensive Care Med. 2010 Jul;36(7):1171-9. doi: 10.1007/s00134-010-1870-0. Epub 2010 Mar 30. PMID 20352189
- [Result] Mahul M, Jung B, Galia F, Molinari N, de Jong A, Coisel Y, Vaschetto R, Matecki S, Chanques G, Brochard L, Jaber S. Spontaneous breathing trial and post-extubation work of breathing in morbidly obese critically ill patients. Crit Care. 2016 Oct 27;20(1):346. doi: 10.1186/s13054-016-1457-4. PMID 27784322